CLINICAL TRIAL: NCT00510419
Title: A Phase 3 Open-Label Study to Assess Subcutaneous Self-Injection With Sumatriptan Succinate Using an Auto-injector During a Single Migraine Attack
Brief Title: A Study to Assess an Auto-injector Being Used to Treat a Migraine Attack
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K644-07-3001
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Migraine
Keywords: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: "Investigational"Auto-injector (sumatriptan succinate)

SUMMARY:
The purpose of this research study is to evaluate an investigational auto-injector system for delivering sumatriptan under the skin for a single migraine attack.

The study could take approximately 5 weeks and will include about 3 office visits to the study doctor, the patient will be contacted every 2 weeks until the patient experiences a migraine and uses the auto-injector. The last visit will be done by a telephone follow-up call.

DETAILED DESCRIPTION:
Investigational Plan:

1. Screening Visit [Visit 0 / 0-14 days prior to receipt of study drug]
2. Baseline Visit [Visit 1 / Provision of study drug and subject training]
3. Treatment Visit [Visit 2 / within 72 hours after study drug administration]
4. Follow-up Visit [Visit 3 / Telephone follow-up 7-10 days after study drug administration]

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 60 years of age
2. Prior effective use of injectable sumatriptan on at least two occasions within the last two months
3. At least two migraines per month suitable injectable sumatriptan
4. Capable of using a migraine self-injection auto-injector
5. Capable of distinguishing between migraine and other headache types (e.g., tension-type headache)

Exclusion Criteria:

1. Seizure disorders
2. Coronary artery disease (CAD)
3. Cardiac dysrhythmia or pacemaker
4. High blood pressure
5. Liver disease
6. Kidney disease
7. Autoimmune disease
8. History of alcohol or substance abuse
9. Currently pregnant
10. Use of any other investigational drug product within 30 days prior to treatment visit

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Successful administration and acceptability of self-injection of sumatriptan under the skin using an investigational auto-injector will be assessed by use of patient-completed scales and a short questionnaire.

SECONDARY OUTCOMES:
• Comparison of pain scores pre-dose and 2 hours post-dose. • Preference of investigational auto-injector experience compared to subject's previous self-administration of sumatriptan.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - San Francisco Clinical Research Center, San Francisco, California
  - New England Center for Headache, Stamford, Connecticut
  - Diamond Head Clinic, Chicago, Illinois
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Clinvest, Springfield, Missouri
  - University of Pittsburgh Headache Center, Pittsburgh, Pennsylvania
  - Wesley Headache Clinic, Memphis, Tennessee
  - Anodyne Headache and Pain Care, Dallas, Texas
  - Houston Headache Clinic, Houston, Texas
  - Road Runner Research, LTD, San Antonio, Texas

REFERENCES:
- [Derived] Landy SH, Tepper SJ, Wein T, Schweizer E, Ramos E. An open-label trial of a sumatriptan auto-injector for migraine in patients currently treated with subcutaneous sumatriptan. Headache. 2013 Jan;53(1):118-125. doi: 10.1111/j.1526-4610.2012.02295.x. Epub 2012 Nov 13. PMID 23148799